CLINICAL TRIAL: NCT00874224
Title: The ORANGE II Trial: An International Multicenter Randomised Controlled Trial of Optimised Surgical Recovery After Left Lateral Hepatic Sectionectomy: Open Versus Laparoscopic Surgery Within an Enhanced Recovery Programme
Brief Title: Surgical Recovery After Left Lateral Hepatic Sectionectomy: Laparoscopic Versus Open Surgery.
Acronym: ORANGE II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); UMC Utrecht (Other); Medisch Spectrum Twente (Other); University Medical Center Groningen (Other); Erasmus Medical Center (Other); University Medical Center Nijmegen (Other); Onze Lieve Vrouwe Gasthuis (Other); Maxima Medical Center (Other); Isala (Other); San Raffaele University Hospital, Italy (Other); University Hospital, Aachen (Other); Deventer Ziekenhuis (Other)
Responsible Party: Principal Investigator, R.S. Fichtinger, Drs. R.M. van dam, Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MEC 08-2-110
Record Dates: First submitted 2009-03-31; First posted 2009-04-02 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Colorectal Cancer; Liver Metastasis; Liver Disease
Keywords: Colorectal cancer liver metastasis; Benign liver disease
MeSH Terms: conditions — Colorectal Neoplasms; Liver Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): patients undergoing open left lateral hepatic sectionectomy
  Interventions: Procedure: open left lateral hepatic sectionectomy
- 2 (Active Comparator): patients undergoing a laparoscopic left lateral hepatic sectionectomy
  Interventions: Procedure: laparoscopic left lateral hepatic sectionectomy
- 3 (Active Comparator): Prospective registry of patients that cannot be randomized (both open and laparoscopic left lateral hepatic sectionectomy)
  Interventions: Procedure: laparoscopic left lateral hepatic sectionectomy; Procedure: open left lateral hepatic sectionectomy

INTERVENTIONS:
Procedure: laparoscopic left lateral hepatic sectionectomy — laparoscopic left lateral hepatic sectionectomy
  Arms: 2; 3
Procedure: open left lateral hepatic sectionectomy — open left lateral hepatic sectionectomy
  Arms: 1; 3

SUMMARY:
The ORANGE II trial is a double blinded randomised controlled trial that will provide evidence on the merits of laparoscopic surgery in patients undergoing a left lateral hepatic sectionectomy in terms of time to functional recovery, hospital length of stay, quality of life, readmission percentage, morbidity and mortality, hospital costs, body image and cosmesis, and long term incidence of incisional hernias.

DETAILED DESCRIPTION:
Recent developments in liver surgery include the introduction of laparoscopic surgery and enhanced recovery programmes. Laparoscopic surgery and enhanced recovery programmes both focus on faster recovery and consequently shorter hospital length of stay.

The ORANGE-II trial is a prospective randomised controlled parallel group superiority trial with a double-blinded experimental and a prospective registry design to determine whether laparoscopic surgery is to be preferred over open surgery in patients undergoing a left lateral hepatic sectionectomy within an enhanced recovery programme. The experimental design produces two randomised arms; (a) open LLS and (b) laparoscopic LLS. An additional registry arm will be based on surgeons/patients that do not want to be randomised because they have an explicit preference for either the laparoscopic LLS or for the open LLS (c).

The primary endpoint of the ORANGE II trial is time to functional recovery. The functional recovery criteria consist of adequate pain control with oral analgetics only, mobility restored to an independent level, absence of intravenous fluid administration, ability to eat solid foods and finally a normal or decreasing serum bilirubin level. A patient is fully functionally recovered when all of the five criteria are satisfied.

Secondary endpoints of this trial are postoperative length of hospital stay, readmission percentage, (liver specific) morbidity, quality of life, body image and cosmetic result, hospital and societal costs during one year and long-term incidence of incisional hernias.

The ORANGE-II trial is a randomised controlled multicentre trial that will provide evidence on the merits of laparoscopic surgery in patients undergoing a left lateral hepatic sectionectomy and participating in an enhanced recovery programme.

ELIGIBILITY:
Inclusion Criteria:

* Patients suitable for undergoing both laparoscopic left lateral sectionectomy as well as open left lateral sectionectomy of the liver.
* Able to understand the nature of the study and what will be required of them.
* Men and non-pregnant, non-lactating women between age 18-80.
* BMI between 18-35.
* Patients with ASA I-II-III

Exclusion Criteria:

* Inability to give written informed consent.
* Patients undergoing liver resection other than left lateral hepatic sectionectomy.
* Patients with ASA IV-V
* Underlying liver disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2010-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Time to functional Recovery | Date the functional recovery criteria are met
  The functional recovery criteria consist of adequate pain control with oral analgetics only, mobility restored to an independent level, absence of intravenous fluid administration, ability to eat solid foods and finally a normal or decreasing serum bilirubin level. A patient is fully functionally recovered when all of the five criteria are satisfied. It is medically justified to discharge patients when the criteria for full functional recovery are met and if the patient is willing to go home.

SECONDARY OUTCOMES:
Postoperative length of hospital stay | 30 days
  including readmission <30 days
Readmission percentage | 1 year
  Readmission percentage during one year follow-up
Total morbidity | 1 year
  Morbidity will be classified and analysed according to the validated classification for postoperative morbidity as described by Dindo et al.
Composite endpoint of liver surgery specific morbidity | 1 year
  Parameter composed of a combination of procedure-specific complications and considered as a single, dichotomous outcome: operative mortality, intra-abdominal haemorrhage, ascites, bile leakage, intra-abdominal abscess and postresectional liver failure. These components, which are all specific to liver surgery and have substantial clinical relevance, reflect Dindo grade 3-5 complications. A composite score of 1 (=failure) will reflect the occurrence of at least one of the above liver specific complications, consequently a score of 0 (=success) will be assigned if none occur.
Quality of life | 1 year
  To assess quality of life the Dutch version of the EQ-5D (EuroQol Group) status test in Dutch centres and the translated EQ-5D for international centres will be used. Furthermore, the EORTC QLQ-C30 with the LM21 module will be used for liver specific treatment measurements. Assessment of the patients' quality of life will be performed at the time of consent, discharge and 10 days, 3, 6 and 12 months after discharge.
Body image and cosmesis | 1 year
  To evaluate differences in postoperative body image and cosmesis, the Body image Questionnaire (BIQ) will be used. The BIQ consists of 8 questions regarding body image and cosmesis. The body image assessment will be performed preoperatively at time of consent. Both the body image and the cosmesis assessment will take place at discharge, 10 days, 3 months, 6 months and 12 months after discharge
Hospital and societal costs | 1 year
  The economic evaluation will include a cost-utility analysis from a Dutch societal perspective. The incremental costs per Quality Adjusted Life Year (QALY) gained will be based on utility scores from the EQ-5D. All hospital expenses (direct and indirect) related to both interventions will be monitored. In addition, a cost questionnaire offered at the regular follow-up consultation (3, 6 and 12 months) will help us to assess the societal and individual costs outside health care relating to patients' absence, impaired mobility, work or normal daily activities.
Incidence of incisional hernias | 1 year
  To assess the incidence of incisional hernias in laparoscopic and open left lateral hepatic sectionectomy patients will be contacted at a mean time of 1 year after resection to receive an ultrasound to diagnose incisional hernia.
Reasons for delay of discharge after functional recovery | untill Discharge
  Factors delaying discharge after functional recovery will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald M van Dam, MD, Study Director — Maastricht University Medical Centre; Cornelis HC Dejong, MD, PhD, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Maastricht University Medical Centre, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Wong-Lun-Hing EM, van Dam RM, van Breukelen GJ, Tanis PJ, Ratti F, van Hillegersberg R, Slooter GD, de Wilt JH, Liem MS, de Boer MT, Klaase JM, Neumann UP, Aldrighetti LA, Dejong CH; ORANGE II Collaborative Group. Randomized clinical trial of open versus laparoscopic left lateral hepatic sectionectomy within an enhanced recovery after surgery programme (ORANGE II study). Br J Surg. 2017 Apr;104(5):525-535. doi: 10.1002/bjs.10438. Epub 2017 Jan 31. PMID 28138958
- [Derived] van Dam RM, Wong-Lun-Hing EM, van Breukelen GJ, Stoot JH, van der Vorst JR, Bemelmans MH, Olde Damink SW, Lassen K, Dejong CH; ORANGE II Study Group. Open versus laparoscopic left lateral hepatic sectionectomy within an enhanced recovery ERAS(R) programme (ORANGE II-trial): study protocol for a randomised controlled trial. Trials. 2012 May 6;13:54. doi: 10.1186/1745-6215-13-54. PMID 22559239